CLINICAL TRIAL: NCT04184557
Title: Effectiveness of a Mindfulness Smartphone App ("Staying Calm in the OR") to Reduce Distress in People With Cancer Waiting for Surgery: A Randomized Controlled Trial
Brief Title: Effectiveness of a Mindfulness Smartphone App to Reduce Emotional Distress in People With Cancer Waiting for Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EC-CS
Record Dates: First submitted 2019-02-12; First posted 2019-12-03 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Cancer
Keywords: cancer; mindfulness; RCT; e-Health; En Calma en el Quirófano; Staying Calm in the OR
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to the intervention arm (app) or to the control arm (treatment as usual [TAU])
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal investigator randomize the participants. Two psychologists who do not know the allocation perform the assessments, mostly through self-reported instruments. Another investigator analyze the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App "Staying Calm in the OR" (Experimental): "Staying Calm in the OR" is a mindfulness-based stress-reduction smartphone tailored for people who are waiting for surgery. It consists of a free, accessible, on-demand, short training through a series of guided meditation practices. They are based on widely studied mindfulness-based programs, such as Mindfulness-Based Stress Reduction (MBSR) or Mindfulness Self Compassion (MSC).
  Interventions: Behavioral: Staying Calm in the OR
- Treatment as Usual (TAU) (No Intervention): Participants assigned to Treatment As Usual (TAU) arm will not download the app until the study is completed.

INTERVENTIONS:
Behavioral: Staying Calm in the OR — "Staying Calm in the OR" is a mindfulness-based stress-reduction smartphone tailored for people who are waiting for surgery. It consists of a free, accessible, on-demand, short training through a series of guided meditation practices. They are based on widely studied mindfulness-based programs, such as Mindfulness-Based Stress Reduction (MBSR) ir Mindfulness Self Compassion (MSC).
  Other Names: En Calma en el Quirófano; EnCalma
  Arms: App "Staying Calm in the OR"

SUMMARY:
Lung cancer and colorectal cancer accounted for the highest number of cancer deceases in 2016. Incidence is around 3.500 cases per year and patients are more commonly men (56%) aged around 69. This study focuses on people with a recent diagnosis of cancer who have been scheduled for surgery.

Evidence suggests that around 11% of people with cancer suffer from anxiety or adjustment disorders and 6,5% hold a diagnosis of major depressive disorder. Moreover, the perioperative period is the most distressing phase of the illness. However, a high number of patients do not have access to mental health services due to either limited resources and geographical limitations or the fear of being stigmatized. The aim is to explore the effectiveness of a mindfulness-based intervention for smartphones designed to reduce pre-surgical distress. It was conceived as a medical tool of prevention), with the purpose of diminishing emotional suffering and clinical complications after surgery. In 2020 Internet will be the most developed technology and almost everyone will have a smartphone; hence, an app for stress reduction will fit in this growing field.

Mindfulness is defined as the ability to pay attention to the present moment with a curious, non-judgmental attitude. Its training consists of both formal meditation practices and informal daily exercises. Mindfulness-based interventions are growing in our National Health System and rigorous researches are being conducted exhibiting good results regarding its effectiveness. However, the fact that Mindfulness instructors must be highly qualified makes these kinds of interventions exceedingly costly to implement. This team is experienced with mindfulness and has developed the app "En Calma en el Quirófano" ("Staying Calm in the OR") to reduce distress before surgery. It consists of a free, accessible, on-demand, short training through a series of guided meditation practices.

In this randomized controlled trial, participants are assigned either to the experimental ("Staying Calm in the OR") or the control arm (treatment as usual). The investigators expect anxiety and depression to be lower in the experimental arm; in addition, the researchers expect that "Staying Calm in the OR" participants will show higher levels of post-surgery recovery.

DETAILED DESCRIPTION:
Lung cancer and colorectal cancer accounted for the highest number of cancer deceases in 2016. Incidence is around 3.500 cases per year and patients are more commonly men (56%) aged around 69. This study focuses on people with a recent diagnosis of cancer who have been scheduled for surgery.

Evidence suggests that around 11% of people with cancer suffer from anxiety or adjustment disorders and 6,5% hold a diagnosis of major depressive disorder. Moreover, the perioperative period is the most distressing phase of the illness. However, a high number of patients do not have access to mental health services due to either limited resources and geographical limitations or the fear of being stigmatized. The aim is to explore the effectiveness of a mindfulness-based intervention for smartphones designed to reduce pre-surgical distress. It was conceived as a medical tool of prevention), with the purpose of diminishing emotional suffering and clinical complications after surgery. In 2020 Internet will be the most developed technology and almost everyone will have a smartphone; hence, an app for stress reduction will fit in this growing field.

Mindfulness is defined as the ability to pay attention to the present moment with a curious, non-judgmental attitude. Its training consists of both formal meditation practices and informal daily exercises. Mindfulness-based interventions are growing in our National Health System and rigorous researches are being conducted exhibiting good results regarding its effectiveness. However, the fact that Mindfulness instructors must be highly qualified makes these kinds of interventions exceedingly costly to implement. This team is experienced with mindfulness and has developed the app "En Calma en el Quirófano" ("Staying Calm in the OR") to reduce distress before surgery. It consists of a free, accessible, on-demand, short training through a series of guided meditation practices.

In this randomized controlled trial, participants are assigned either to the experimental ("Staying Calm in the OR") or the control arm (treatment as usual). The investigators expect anxiety and depression to be lower in the experimental arm; in addition, the researchers expect that EnCalma participants will show higher levels of post-surgery recovery.

Main hypothesis. Anxiety and depression symptoms will be significantly lower in the experimental arm after Staying Calm in the OR" training.

Secondary hypotheses. Recovery after surgery will be higher amongst participants in the experimental arm, who will exhibit fewer post-surgical complications, lower rates of hospitalizations, lower levels of analgesia, shorter hospitalizations and a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 100 years old
* Diagnosis of cancer
* Being in waitlist for surgery for less than 14 days
* Signed informed consent

Exclusion Criteria:

* Acute severe mental disorder according to DSM-5 diagnostic criteria
* Not having a smartphone
* Not being able to download and use the smartphone app "Calm before Surgery"

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in anxiety and depression | From baseline (15 days before surgery) to hospital discharge (around 7 days after surgery)
  Change in Hospital Anxiety and Depression Scale (HADS). Anxiety and depressive symptoms are measured with this self-reported instrument. The scores of the 15 items range from 0 to 4. The final score is the summatory of these items and range from 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

SECONDARY OUTCOMES:
Change in quality of life | From baseline (15 days before surgery) to hospital discharge (around 7 days after surgery)
  Change in World Health Organization Quality of Life Brief Scale (WHOQOL-BREF). This is a self-reported instrument that how much the person is satisfied with many aspects of his or her live, and general domains of the quality of life construct. There are 26 items and each one is scored from 0 to 5. Higher scores suggest better quality of life in direct items and poorer quality of life in reverse items. The final score range from 0 to 130, and the higher the score the better the perceived quality of life.
Change in pain experience | From baseline (15 days before surgery) to hospital discharge (around 7 days after surgery)
  Change in Visual Analog Scale (VAS) for pain. In this visual scale, the evaluator needs to rate how much pain is he or she experiencing in the present moment. Scores range from 0 (no pain at all) to 10 (extreme pain).
Presence of post-surgery complications | Clavien-Dindo Scale score at hospital discharge (around 7 days after surgery)
  Clavien-Dindo Scale score. This scale measures complications in surgery. They evaluator has to choose among the following categories:
  Grade I. Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. This grade also includes wound infections opened at the bedside.
  Grade II. Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusions and total parenteral nutrition also included.
  Grade III. Requiring surgical, endoscopic or radiological intervention
  * IIIa. Intervention not under general anesthesia
  * IIIb. Intervention under general anesthesia
  Grade IV. Life-threatening complication (including CNS complications) requiring IC/ICU-management
  * IVa. Single organ dysfunction (including dialysis)
  * IVb. Multiple organ dysfunction
  Grade V Death of a patient
Change in blood pressure | From surgery to hospital discharge (around 7 days after surgery)
  Change in blood pressure, as registered by nursers during the hospitalization period
Change in oxygen saturation | From surgery to hospital discharge (around 7 days after surgery)
  Change in oxygen saturation, as registered by nursers during the hospitalization period
Change in temperature | From surgery to hospital discharge (around 7 days after surgery)
  Change in temperature, as registered by nursers during the hospitalization period
Change in analgesia | From surgery to hospital discharge (around 7 days after surgery)
  Change in analgesia, as registered by nursers during the hospitalization period

OTHER OUTCOMES:
Level of satisfaction with "Calm Before Surgery" | Hospital discharge (around 7 days after surgery)
  Level of satisfaction with smartphone app "Calm Before Surgery" measured by Client Satisfaction Questionnaire (CSQ-8). This 8-item instrument explores how much a person is satisfied with different domains of healthcare services. A final score between 8 and 32 is provided, with higher values indicating higher levels of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodríguez-Vega, PhD, Principal Investigator — La Paz University Hospital; Madrid Autonomous University
Locations (2):
- Spain (2):
  - 12 Octubre University Hospital, Madrid
  - La Paz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available one year after publishing the final results for at least 5 years
Access Criteria: Please contact PI Beatriz Rodríguez-Vega (beatrizrvega@gmail.com)

REFERENCES:
- See also: Download "En Calma en el Quirófano" for iOS — https://itunes.apple.com/sc/app/en-calma-en-el-quirófano/id1244782979?mt=8
- See also: Download "En Calma en el Quirófano" for Android — https://play.google.com/store/apps/details?id=es.sw.mindfulness&hl=es